CLINICAL TRIAL: NCT03246178
Title: A Research on Haploidentical Transplantation in Severe Aplastic Anemia Using Reduced-intensity Fludarabine-based Conditioning
Brief Title: Haploidentical Transplantation in Severe Aplastic Anemia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Wu Xiaoxiong (Other)
Responsible Party: Sponsor-Investigator, Wu Xiaoxiong, Head, Research group of the Center of Hematology, Chinese PLA General Hospital
Organization: Chinese PLA General Hospital (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2016QX-KS008
Record Dates: First submitted 2017-05-01; First posted 2017-08-11 (Actual); Last update posted 2017-08-11 (Actual); Status verified 2017-08

CONDITIONS: Severe Aplastic Anemia
Keywords: Haploidentical; Hematopoietic stem cell transplantation; Severe aplastic anemia
MeSH Terms: conditions — Anemia, Aplastic

STUDY DESIGN:
Intervention Model Description: Patients with SAA
Masking Description: no masking
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MSD-HSCT (Other): This group received treatment of matched sibling donor - hematopoietic stem cell transplantation (MSD-HSCT).
  Interventions: Other: MSD-HSCT
- HFD-HSCT (Experimental): This group received treatment of haploid family donor - hematopoietic stem cell transplantation (HFD-HSCT).
  Interventions: Other: HFD-HSCT

INTERVENTIONS:
Other: MSD-HSCT — 1. Conditioning regimens: (A) Patients had SAA and PNH, or heavy transfusion (RBC≥25U), or failed rabbit ATG therapy, and received 0.8 mg/kg/6h busulfan (days -7 to -6), 30mg/m2/day fludarabine (days -5 to -2), 25 mg/kg/day cyclophosphamide (days -5 to -2) and 2.5 mg/kg/day r-ATG (days -5 to -2). (B) The other patients with SAA or VSAA received same procedure but without busulfan;
  2. Allogeneic HSC infusion: Doner BM cells were harvested to achieve a target mononuclear cell count (MNC) of 2-4 × 108 per kilogram of recipient weight. The target MNC from PB was 4-6× 108 per kilogram of recipient weight;
  3. Prophylaxis and treatment of GVHD: GVHD prophylaxis consisted of intravenous CSP 2-3 mg/kg/day in divided doses beginning on the day before transplantation (day -5) and the target concentration was adjusted to 150-250 ng/ml. The oral MMF dose was 20 mg/kg/day from day -1 and was tapered off after 1 months if no aGVHD was observed.
  Arms: MSD-HSCT
Other: HFD-HSCT — 1. Conditioning regimens: (A) Patients had SAA and PNH, or heavy transfusion (RBC≥25U), or failed rabbit ATG therapy, and received 0.8 mg/kg/6h busulfan (days -7 to -6), 35mg/m2/day fludarabine (days -5 to -2), 25 mg/kg/day cyclophosphamide (days -5 to -2) and 2.5 mg/kg/day r-ATG (days -5 to -2). (B) The other patients with SAA or VSAA received same procedure but without busulfan;
  2. Allogeneic HSC infusion: Doner BM cells were harvested to achieve a target mononuclear cell count (MNC) of 2-4 × 108 per kilogram of recipient weight. The target MNC from PB was 4-6× 108 per kilogram of recipient weight;
  3. Prophylaxis and treatment of GVHD: GVHD prophylaxis consisted of intravenous CSP 2-3 mg/kg/day in divided doses beginning on the day before transplantation (day -5) and the target concentration was adjusted to 200-300 ng/ml. The oral MMF dose was 20 mg/kg/day from day -3 and was tapered off after 2 months if no aGVHD was observed.
  Arms: HFD-HSCT

SUMMARY:
This is a prospective case-control study on SAA patients treated with HSCT, order to further discuss and assess the safety, feasibility and effectiveness of HFD-HSCT which performed with reduced-intensity fludarabine-based conditioning regimen.Our findings would indicate that SAA patients who lack MSD benefited most if HFD-HSCT was performed with reduced-intensity fludarabine-based conditioning regimen, and our improved outcomes with HFD-HSCT may lead to a salvaged therapy and an expanded direct role for SAA in the future.

ELIGIBILITY:
Inclusion Criteria:

(i) Diagnosis of SAA, very SAA or SAA and paroxysmal nocturnal hemoglobinuria (PNH) according to the International Aplastic Anemia Study Group; (ii) SAA patients no response to previous IST; (iii) adequate performance status [Eastern Cooperative Oncology Group (ECOG) score 0-2].

Exclusion Criteria:

(i) Congenital forms of aplastic anemia; (ii)Patients with any severe pulmonary, cardiac, liver, or renal diseases or active infection.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2017-07-10 (Actual); Primary Completion 2020-07-01 (Estimated); Study Completion 2020-12-01 (Estimated)

PRIMARY OUTCOMES:
Engraftment | In the first months after infusion
  Neutrophil engraftment was defined as the first of three consecutive days in which the neutrophil counts (ANC) exceeded 0.50 × 109/L, and platelet engraftment was defined as the first of five consecutive days in which the platelet count exceeded 20 × 109/L without transfusion. GF was classified as follows: (1) primary non-engraftment (failure to reach a neutrophil count of 0.5×109/L after transplant); (2) rejection (decrease in blood counts to < 0.5×109/L neutrophils, after achieving a neutrophil count of 0.5×109/L); (3) late graft failure (decrease of blood counts after day 100 to < 1.0×109/L neutrophils and < 30×109/L platelets).
Toxicity grading | TRT was defined as toxic effects occurring within 40 days after HSCT
  The transplantation-related toxicity (TRT) was graded using the National Cancer Institute Common Toxicity Criteria for Adverse Events version 4.0. Organ damage due to GVHD or infectious complications were excluded.
Chimerism analyses +30 | Days +30 after HSCT
  Chimerism would be evaluated in recipient BM cells usually on days +30 after HSCT using cytogenetic G-banding or fluorescence in situ hybridization. Sex-matched donor-recipient chimerism was assessed using PCR-based analyses of polymorphic minisatellite or microsatellite regions. HLA typing was performed for patients with HLA-haploidentical donors.
Chimerism analyses +100 | Days +100 after HSCT
  Chimerism would be evaluated in recipient BM cells usually on days +180 after HSCT using cytogenetic G-banding or fluorescence in situ hybridization. Sex-matched donor-recipient chimerism was assessed using PCR-based analyses of polymorphic minisatellite or microsatellite regions. HLA typing was performed for patients with HLA-haploidentical donors.
Chimerism analyses +180 | Days +180 after HSCT
  Chimerism would be evaluated in recipient BM cells usually on days +100 after HSCT using cytogenetic G-banding or fluorescence in situ hybridization. Sex-matched donor-recipient chimerism was assessed using PCR-based analyses of polymorphic minisatellite or microsatellite regions. HLA typing was performed for patients with HLA-haploidentical donors.
Chimerism analyses +365 | Days +365 after HSCT
  Chimerism would be evaluated in recipient BM cells usually on days +365 after HSCT using cytogenetic G-banding or fluorescence in situ hybridization. Sex-matched donor-recipient chimerism was assessed using PCR-based analyses of polymorphic minisatellite or microsatellite regions. HLA typing was performed for patients with HLA-haploidentical donors.
OS 1-year | 1-year after HSCT
  OS was defined as the time from transplantation to death from any cause or the last follow-up.
OS 2-year | 2-year after HSCT
  OS was defined as the time from transplantation to death from any cause or the last follow-up.
OS 5-year | 5-year after HSCT
  OS was defined as the time from transplantation to death from any cause or the last follow-up.
EFS 1-year | 1-year after HSCT
  EFS was defined as survival with a response to therapy. Death, GF and relapse were considered as treatment failure.
  EFS was defined as survival with a response to therapy. Death, GF and relapse were considered as treatment failure.
EFS 2-year | 2-year after HSCT
  EFS was defined as survival with a response to therapy. Death, GF and relapse were considered as treatment failure.
EFS 5-year | 5-year after HSCT
  EFS was defined as survival with a response to therapy. Death, GF and relapse were considered as treatment failure.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoxiong WU, PhD, Study Director — The First Affiliated Hospital of General Hospital of PLA
Locations (1):
- Department of Hematology, 304th Clinical Division, Chinese PLA General Hospital, Beijing, China